CLINICAL TRIAL: NCT06017271
Title: Predictive Value of Epicardial Adipose Tissue for Pulmonary Embolism and Death in Patients With Lung Cancer
Status: Withdrawn | Type: Observational
Why Stopped: The number of patients is not sufficient to support the project.
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2023LSK-269
Record Dates: First submitted 2023-08-24; First posted 2023-08-30 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Pulmonary Embolism; Lung Cancer
MeSH Terms: conditions — Pulmonary Embolism; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PE group: The CTPA diagnosis suggest pulmonary embolism
  Interventions: Diagnostic Test: CTPA (computed tomography pulmonary angiography)
- control group: The CTPA diagnosis did not suggest pulmonary embolism
  Interventions: Diagnostic Test: CTPA (computed tomography pulmonary angiography)

INTERVENTIONS:
Diagnostic Test: CTPA (computed tomography pulmonary angiography) — The CTPA diagnosis suggest or did not suggest pulmonary embolism.

SUMMARY:
The occurrence and progression of lung cancer is related to visceral adipose tissue (VAT). Epicardial adipose tissue (EAT) is a kind of VAT, producing a variety of inflammatory cytokines and adipokines, participating in the formation of local inflammation, promoting the formation of pre-thrombotic state, and leading to the occurrence of thromboembolism. Patients with lung cancer have increased inflammatory response and are more prone to suffer thrombosis. However, in lung cancer patients, the clinical correlation between EAT and pulmonary embolism has not been reported. Objective: To analyze the risk factors of poor prognosis in lung cancer patients with PE, and to explore the predictive value of EAT in pulmonary embolism events and death in lung cancer patients. Methods: EAT volume and density, as well as anthropometric and blood biomarkers, were evaluated in a sample of lung cancer patients, half with pulmonary embolism and half without. The incidence of adverse prognosis and related factors were followed up by telephone.

ELIGIBILITY:
Inclusion Criteria:

* The pathological diagnosis was lung cancer
* Pulmonary artery was evaluated by CTA during hospitalization.

Exclusion Criteria:

* Patients with incomplete clinical data
* Patients with no follow-up data
* Patients with a history of PE before diagnosis of lung cancer

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study was conducted on patients with a confirmed diagnosis of Lung Cancer who were admitted to the First Affiliated Hospital of Xi'an Jiaotong University from 1 January 2012 to 31 December 2021. Patients who did not meet any of the inclusion criteria or met any of the exclusion criteria were excluded. The subjects were divided into PE group and control group according to the results of CTPA examination, and the patients in the two groups were matched by gender and age 1:1 tendency score.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-19 (Actual)

PRIMARY OUTCOMES:
EAT volume | May, 20, 2023
  volume of epicardial adipose tissue (EAT), Cm3
EAT density | May, 20, 2023
  density of epicardial adipose tissue (EAT) , Hounsfield Units (HU)

CONTACTS AND LOCATIONS:
Overall Officials: Yang Yan, Study Director — First Affiliated Hospital Xi'an Jiaotong University; Haichen Wang, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided